CLINICAL TRIAL: NCT01805531
Title: Satisfaction and Quality of Life in Patients With a Diagnosis of Non Valvular Atrial Fibrillation Who Take Rivaroxaban for Stroke Prevention
Brief Title: Satisfaction/Quality of Life With Rivaroxaban in SPAF (Stroke Prevention in Atrial Fibrillation) Indication
Acronym: SAFARI
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 16398; XA1213FR (Other: Company internal)
Record Dates: First submitted 2013-03-05; First posted 2013-03-06 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Atrial Fibrillation
Keywords: SF36 questionnaire; Anti Clot Treatment Scale; Satisfaction; Quality of Life; Rivaroxaban; Stroke prevention
MeSH Terms: conditions — Atrial Fibrillation; Personal Satisfaction | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rivaroxaban
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — 20 mg po once daily, which is also the recommended maximum dose. In subjects with moderate creatinine clearance (30-49 ml/min), the dose 15 mg once daily is recommended.

SUMMARY:
National, multicenter, prospective, observational, non-interventional study. The objective is to determine if the switch from Vitamin K antagonists (VKA) to Xarelto in subjects treated with VKA with issues for stroke prevention in non valvular atrial fibrillation is associated with an improvement of the treatment satisfaction after 3 months. The treatment satisfaction will be measured by the Anti Clot Treatment Scale (ACTS) score.

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects ≥ 18 years of age with a diagnosis of non-valvular atrial fibrillation
* Who are treated with Vitamin K antagonists (VKA) with issues for at least the 4 previous weeks (issues are assessed on medical judgment)
* Who start treatment with rivaroxaban to prevent stroke or non-CNS (central nervous system) systemic embolism
* With anticoagulation therapy planned for at least 6 months

Exclusion Criteria:

* Contra indication to the use of Xarelto as described in the Summary of Product Characteristics (SmPC); key contra indications are:

  * Hypersensitivity to the active substance or to any of the excipients listed in SmPC section 6.1.
  * Lesion or condition at significant risk of major bleeding
  * Concomitant treatment with any other anticoagulant agent
  * Clinically significant active bleeding
  * Hepatic disease associated with coagulopathy and clinically relevant bleeding risk including cirrhotic patients with Child Pugh B and C
  * Pregnancy and breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients more than 18 years old, with a diagnosis of non-valvular atrial fibrillation, treated to prevent stroke or non-central nervous system systemic embolism, who switch from VKA to Xarelto due to issues with VKA
Sampling Method: Non-Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change of the Anti Clot Treatment Scale (ACTS) score at 3 months compared with baseline score | After 3 months

SECONDARY OUTCOMES:
Change of ACTS score after 1 and 6 months of treatment | After 1 and 6 months
Continuation rate at 1, 3 and 6 months | After 1, 3 and 6 months
Change of SF36 score at 1, 3 and 6 months (health related quality of life determined by SF36 questionnaire) | After 1, 3 and 6 months
Physician's satisfaction at 1, 3 and 6 months assessed by a 5-point Likert scale response ("very satisfied", "satisfied", "neutral", "unsatisfied" or "very unsatisfied") | After 1, 3 and 6 months
Patient's compliance with VKA treatment at baseline and with Xarelto treatment at 1, 3 and 6 months assessed by the investigator as good (≥80%), average (50-80%) or poor (<50%) | After 1, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, France